CLINICAL TRIAL: NCT07031076
Title: Investigating the Cognitive and Brain Health Benefits of Lean Pork Consumption
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigative team has transferred to another university.
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: National Pork Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 23280
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Dietary Intervention; Dietary Proteins; Dietary Assessment; Older Adults (65 Years and Older); Cognitive Ability, General
Keywords: pork consumption; pork dietary intervention; brain health; cognitive health
MeSH Terms: interventions — Freezing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will participate in the 16-week lean pork dietary intervention study. Participants will be provided with 4 portions of ready-to-eat lean pork in frozen packages per week. Each portion of ready-to-eat lean pork provided to this group will weigh 5 ounces.
  Interventions: Dietary Supplement: Ready-to-eat lean pork in frozen, 5-oz packages
- Control Group (No Intervention): The control group will not participate in any dietary intervention, other than being instructed to maintain their regular diet.

INTERVENTIONS:
Dietary Supplement: Ready-to-eat lean pork in frozen, 5-oz packages — The dietary intervention lasts 16 weeks for each individual. Participants in the experimental group will receive this intervention. Each participant will acquire 4 portions of ready-to eat lean pork in frozen packages per week; each portion of ready-to-eat lean pork in this intervention will weigh 5 ounces.
  Arms: Experimental Group

SUMMARY:
The goal of this clinical trial is to learn if eating more lean pork will lead to better cognition and a healthier brain in older adults. The main questions it aims to answer are:

* Does eating more lean pork lead to higher scores on cognitive tests and better quality of life?
* Does eating more lean pork lead to slower brain aging and/or better brain function?

Researchers will compare participants in the experimental group (participants undergoing the dietary intervention) to control participants (participants that do not undergo the intervention).

Participants will:

* Be instructed to prepare and consume ready-to-eat pork meals along with their regular diet and not eat any more pork other than what they are given; or be instructed to consume their regular diet
* Visit the study facilities once every week to pick up ready-to-eat pork meals and complete dietary surveys; or complete dietary surveys every 4 weeks
* Visit the study facilities before and after the 16-week of intervention period for researchers to study them

DETAILED DESCRIPTION:
The goal of this study is to evaluate the effects of learn pork consumption on cognitive and brain health in healthy older adults. Specifically, we seek to evaluate the effects of lean pork consumption on measures of executive function, memory, psychological well-being, and sleep quality. Additionally, we will explore the effects of increased lean pork consumption on measures of brain health derived from structural and functional brain imaging.

The study will consist of two groups of participants: experimental and control. Participants in the experimental group will take part in a 16-week dietary intervention. Throughout the intervention, participants in the experimental group will receive 4 portions of ready-to-eat lean pork in frozen packages each week. Each serving of ready-to-eat lean pork for the experimental group will weigh 5-ounces. Participants in the control group will be asked to continue their regular diet, without receiving any frozen packages of ready-to-eat lean pork. Study compliance will be evaluated through weekly surveys about lean pork consumption.

In addition, all participants will complete pre- and post-intervention assessments:

* MRI scan, including structural and functional brain imaging
* a comprehensive questionnaire battery evaluating cognitive and psychological measures
* neuropsychological tasks
* a blood draw

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study
* Males and females; Age 65-75
* Willingness to adhere to the ready-to-eat lean pork intervention regimen or the control condition regimen (depending on group assignment)
* Score between 51 and 80 out of 100 on the Healthy Eating Index
* Consume less than or equal to 15 grams of lean pork per day on average prior to participating in the study
* BMI between 18.5 and 39.9
* Mini-Mental State Examination score 26 or greater
* Vision scored greater than 20/50
* No history of subjective cognitive impairment
* No evidence of loss of instrumental activities of daily living
* Minimal dependence in hygiene, bathing, and dressing
* Low pork consumers
* Willing to discontinue dietary supplement use throughout the duration of the study, if they are consuming supplement at the time of the registration
* No known contraindication to MRI scans as determined by the MRI screening survey questions

Exclusion Criteria:

* Current use of medications that may affect their responses to dietary intervention, such as amphetamines, antidepressants, anti-diabetic medications, laxatives, antibiotics, statins and diuretics.
* Known intolerance or allergy to pork
* Current use of nicotine products, including vaping
* Previous use of nicotine products, including vaping, within the recent 6 months at the time of pre-screening
* Diagnosis of mild cognitive impairment
* Diagnosis of any dementia, including, but not limited to, Alzheimer's Disease, Lewy body disease, vascular cognitive impairment and frontotemporal dementia
* Diagnosis of psychiatric illness within the last 3 years
* Stroke in previous 12 months
* Cancer diagnosis within past 3 years, except prostate cancer or basal cell carcinoma
* Current chemotherapy or radiation treatment
* Planned move from study area
* Scheduling conflicts that would preclude participation in study activities
* Prior or ongoing involvement in cognitive training or dietary intervention studies
* Contraindications for MRI
* Dietary quality outside the average range (i.e., HEI score less than 51 or greater than 80)
* Other inability to complete study activities

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
WAIS-V | Baseline and after 16 weeks
  Wechsler Adult Intelligence Scale, verison 5. Comprehensive assessment battery for measuring cognitive abilities
Trail Making Test | Baseline and after 16 weeks
  Delis-Kaplan Executive Function System test for sequencing and cognitive flexibility
NIH Toolbox (Dimensional Change Card Sort) | Baseline and after 16 weeks
  Test for executive function and cognitive flexibility
NIH Toolbox (Flanker) | Baseline and after 16 weeks
  test for executive functions: attention and inhibitory control
NIH Toolbox (List Sorting Working Memory Test) | Baseline and after 16 weeks
  Test for working memory
Adult Decision-Making Competence test | Baseline and after 16 weeks
  Assessment of how well adults make decisions. Subcategories include Resistance to Framing, Recognizing Social Norms, Under/Overconfidence, Applying Decision Rules, Consistency in Risk Perception, and Resistance to Sunk Costs
Cognitive Reflection Test | Baseline and after 16 weeks
  Test to measure the ability to suppress an intuitive wrong answer in favor of a more reflective correct answer
Attentional Network Task | Baseline and after 16 weeks
  Computerized task to measure the effects of visual and auditory cues on visual processing
UCLA Loneliness Scale | Baseline and after 16 weeks
  measure of subjective loneliness and social isolation
Short Form-36 Health Survey | Baseline and after 16 weeks
  self-report measure of health status and quality of life
Psychological Wellbeing Scale | Baseline and after 16 weeks
  the psychological wellbeing scale assesses six aspects of psychological wellbeing and happiness: Autonomy, Environmental Mastery, Personal Growth, Positive Relations with Others, Purpose in Life, Self-Acceptance
Decision Outcome Inventory | Baseline and after 16 weeks
  an assessment of outcomes of real-life decisions
The Mindset Survey | Baseline and after 16 weeks
  an assessment to determine whether an individual has a fixed mindset or a growth mindset
Need for Cognition Scale | Baseline and after 16 weeks
  assessment of an individual's tendency to engage in and enjoy thinking or mental exertion
Pittsburgh Sleep Quality Index | Baseline and after 16 weeks
  Self-report assessment of sleep quality over the past month. The survey includes measures related to Sleep Latency, Sleep Duration, Sleep Efficiency, Sleep Disturbances, Use of Sleep Medications, Daytime Fatigue, and Sleep Quality
Consortium to Establish a Registry for Alzhiemer's Disease Word List Acquisition and Delayed Recall | Baseline and after 16 weeks
  A learning and delay memory recall task that is used to quickly assess an individual's mental capacity in memory.
Geriatric Depression Scale | Baseline and after 16 weeks
  Assessment of an older adult's status of mental health that screens for depression
Ohio State Traumatic Brain Injury Identification | Baseline and after 16 weeks
  Interview-style assessment of past head injuries, including their severity and their resulting symptoms.
Symptom Checklist 90-Revised | Baseline and after 16 weeks
  self-report assessment of psychological symptoms related to the domains of somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism
Grit | Baseline and after 16 weeks
  self-report measure of perseverance
Brief Dispositional Resilience Scale | Baseline and after 16 weeks
  a 15-item measure of psychological hardiness, covering aspects related to commitment, control, and challenge
Valence Bias Task | Baseline and after 16 weeks
  an assessment to measure an individual's tendency to interpret ambiguous stimuli as having a positive or negative valence

SECONDARY OUTCOMES:
Brain Imaging | Baseline and after 16 weeks
  * T1- and T2-weighted imaging to visualize the structure of the brain
  * Functional MRI of the whole brain to examine changes in brain activity and functional topology
  * Diffusion tensor imaging to map the white matter structures in the brain
  * Magnetic resonance elastography to examine the elasticity of brain tissues
  * Susceptibility weighted imaging to examine cerebrovascular health

OTHER OUTCOMES:
Height | Baseline and after 16 weeks
  measured in feet and inches
Weight | Baseline and after 16 weeks
  measured in pounds (lbs)
Body Mass Index | Baseline and after 16 weeks
  Calculated by body mass divided by the square of the body height, unit in kg/m^2
Heart Rate | Baseline and after 16 weeks
  Heart rate will be measured over 5-minute intervals, when the participants are sitting up right on a chair without any physical exhaustion condition. Heart rate will be reported as beat per minute by averaging the heart activity over the 5-minute intervals.
Heart Rate Variability | Baseline and after 16 weeks
  Heart rate variability will be measured as the standard deviation of R-R interval in millisecond as unit.
Systolic and diastolic Blood Pressure | Baseline and after 16 weeks
  Measured in mmHg
Body Composition | Baseline and after 16 weeks
  Body composition will be measured in body fat%, using a bioimpedance scale
Grip Strength | Baseline and after 16 weeks
  Participants will squeeze a hydraulic device three times with their right hand. Grip strength will be obtained by averaging the three measurements, which will be measured in kilograms.
Blood-based biomarkers associated with consumption of lean pork | Baseline and after 16 weeks
  Biomarkers under evaluation include inflammatory biomarkers and nutrient biomarkers in blood from participants in the experimental group

CONTACTS AND LOCATIONS:
Overall Officials: Aron Barbey, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- University of Nebraska-Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Study findings will be submitted to peer-reviewed journals such as those that follow the ICMJE's recommendations for the Conduct, Reporting, Editing and Publication of Scholarly Work in Medical Journals. The data collected during this project may be shared through public-use files, repositories or other means outside of the approved research team as a requirement of publication. All data will be identified with subject IDs only when shared. Research records such as informed consent forms, MRI Safety Screening forms, research compliance records, masterlist linking names to subject IDs will not be shared.
Supporting Information: Study Protocol, Analytic Code
Time Frame: IPD and supporting information will be available beginning 1 year after the publication of results with no end date.
Access Criteria: Researchers who provide a methodologically sound proposal will be able to access the IPD and supporting information. Researchers are not restricted on the type of analyses, as long as they are methodologically sound. The statistical methods for those analyses must be approved before the researchers can gain access to the data.
  For data sharing, a proposal that describes planned analyses must be submitted to the study's contact personnel for review. A data sharing agreement must be signed between the institution of the requesting researchers and the institution of the study's principal investigator.

REFERENCES:
- [Background] Wade AT, Davis CR, Dyer KA, Hodgson JM, Woodman RJ, Keage HAD, Murphy KJ. A Mediterranean Diet with Fresh, Lean Pork Improves Processing Speed and Mood: Cognitive Findings from the MedPork Randomised Controlled Trial. Nutrients. 2019 Jul 4;11(7):1521. doi: 10.3390/nu11071521. PMID 31277446
- [Background] Hepsomali P, Groeger JA. Diet and general cognitive ability in the UK Biobank dataset. Sci Rep. 2021 Jun 3;11(1):11786. doi: 10.1038/s41598-021-91259-3. PMID 34083695
- [Background] Zhang H, Hardie L, Bawajeeh AO, Cade J. Meat Consumption, Cognitive Function and Disorders: A Systematic Review with Narrative Synthesis and Meta-Analysis. Nutrients. 2020 May 24;12(5):1528. doi: 10.3390/nu12051528. PMID 32456281